CLINICAL TRIAL: NCT03644797
Title: Second Molecular Event Identification by Exome Sequencing for Intellectually Disabled Patients Carrying 16p13.11 CNVs
Acronym: SEESIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0693
Record Dates: First submitted 2018-07-05; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients presenting intellectual disability and previously diagnosed as carriers of a 16p13.11 copy number variant using Cytogenetic Micro Array.
  Interventions: Genetic: Exome sequencing

INTERVENTIONS:
Genetic: Exome sequencing — Detection of a second (likely) pathogenic molecular event on exome data for intellectual disability beyond the 16p13.11 Copy Number Variant.

SUMMARY:
16p13.11 copy number variations are considered as predisposition factors for neurodevelopmental disorders but can be inherited from normal parents. SEESIC aims at identifying seond molecular events by exome sequencing that could modulate the phenotype and explain familial discrepancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting intellectual disability
* Patients carrying a 16p13.11 copy number variant
* Blood DNA available without re sampling for the patient and his parents.
* Consent for genetics analysis already for the patient and his parents.

Exclusion Criteria:

- Other diagnosis for intellectual disability (apart 16p13.11 copy number variant) already posed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting intellectual disability and carrying a 16p13.11 copy number variant.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Second pathogenic molecular event on exome data | 4 months
  Number of participants diagnosed as carrier of a (likely) pathogenic variation beyond 16p13.11 CNV through exome sequencing according to ACMG 2015 guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CHATRON, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant (Groupement Hospitalier Est), Bron, France